CLINICAL TRIAL: NCT01529034
Title: An Open-Label Safety Study of USL261 in the Outpatient Treatment of Subjects With Seizure Clusters
Brief Title: Study to Evaluate the Long-term Safety and Tolerability of USL261 in Patients With Seizure Clusters
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P261-402; 2011-004109-25 (EudraCT Number)
Record Dates: First submitted 2012-02-03; First posted 2012-02-08 (Estimated); Results first posted 2019-06-25 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Epilepsy
Keywords: Epilepsy; seizure clusters; acute repetitive seizures; rescue treatment
MeSH Terms: conditions — Epilepsy

ARMS (1):
- USL261 (Experimental): Intranasal midazolam 5 mg
  Interventions: Drug: USL261

INTERVENTIONS:
Drug: USL261

SUMMARY:
The purpose of this study is to examine the long-term safety and tolerability of USL261 in the treatment of seizure clusters.

DETAILED DESCRIPTION:
Participants who completed study P261-401 (NCT01390220), a randomized double-blind study of USL261 (intranasal midazolam) versus placebo to acutely treat a seizure cluster episode, were eligible to to enroll in this open-label extension study (P261-402). The participant's caregiver administered a USL261 5 milligram (mg) dose for a seizure episode meeting study criteria. A second USL261 5 mg dose could be administered after 10 minutes and up to 6 hours after the first dose for persistent or recurrent seizures, unless the participant met exclusions to administration of the second dose. A participant could have more than 1 seizure cluster episode treated during his/her study participation.

ELIGIBILITY:
Inclusion Criteria:

* Has a competent, adult caregiver who can recognize and observe the subject's seizure cluster episodes
* Has successfully completed study P261-401, and the subject and caregiver have demonstrated adequate compliance with P261-401 study procedures as determined by the investigator

Exclusion Criteria:

* Has experienced status epilepticus during or since the P261-401 study
* In the opinion of the investigator, is experiencing an ongoing, uncontrolled, clinically significant adverse event(s) from P261-401 at Visit 1 or did experience a clinically significant adverse event in study P261-401 that might prevent the subject from safely participating in the study
* Has a neurological disorder that is likely to progress in the next year
* Has a history of acute narrow-angle glaucoma
* Has a medical condition including uncontrolled cardiac, pulmonary, renal, hepatic, or gastrointestinal disease that could interfere with the study, subject safety/safety monitoring, or is not stable despite current therapy
* Subject has severe chronic cardio-respiratory disease or the need for ambulatory oxygen
* Has had psychogenic, non-epileptic seizure(s) during or since the P261-401 study
* Has active suicidal plan or intent as determined by the C-SSRS at Visit 1 or medical history
* Subject has had vagus nerve stimulator (VNS) implanted since the completion of study P261-401

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (58):
- United States (31):
  - United States, Arizona, Phoenix, Arizona
  - United States, Arizona, Scottsdale, Arizona
  - United States, Arizona, Tucson, Arizona
  - United States, Arkansas, Little Rock, Arkansas
  - United States, California, Fresno, California
  - United States, California, Sacramento, California
  - United States, California, Ventura, California
  - United States, Colorado, Aurora, Colorado
  - United States, Connecticut, New Haven, Connecticut
  - United States, Florida, Port Charlotte, Florida
  - United States, Florida, Wellington, Florida
  - United States, Idaho, Boise, Idaho
  - United States, Illinois, Chicago, Illinois
  - United States, Kentucky, Lexington, Kentucky
  - United States, Maryland, Baltimore, Maryland
  - United States, Michigan, Detroit, Michigan
  - United States, Minnesota, Saint Paul, Minnesota
  - United States, Missouri, St Louis, Missouri
  - United States, New Hampshire, Lebanon, New Hampshire
  - United States, New Jersey, Hackensack, New Jersey
  - United States, New York, New York, New York
  - United States, New York, Stony Brook, New York
  - United States, New York, The Bronx, New York
  - United States, North Carolina, Durham, North Carolina
  - United States, North Carolina, Winston-Salem, North Carolina
  - United States, Oklahoma, Oklahoma City, Oklahoma
  - United States, Pennsylvania, Philadelphia, Pennsylvania
  - United States, Tennessee, Memphis, Tennessee
  - United States, Tennessee, Nashville, Tennessee
  - United States, Texas, Dallas, Texas
  - United States, Texas, Greenville, Texas
- Australia (3):
  - Australia, New South Wales, Randwick, New South Wales
  - Australia, Victoria, Heidelberg West, Victoria
  - Australia, Victoria, Parkville, Victoria
- Canada (3):
  - Canada, Montreal, Ontario
  - Canada, Toronto, Toronto, Ontario
  - Canada, Toronto, Quebec
- Germany (4):
  - Germany, München, Bavaria
  - Germany, Marberg, Hesse
  - Germany, Bonn, North Rhine-Westphalia
  - Germany, Bielefeld, Westfalen-Lippe
- Hungary, Budapest, Hungary
- Israel (3):
  - Israel, Haifa
  - Israel, Petah Tikvah
  - Israel, Ramat Gan
- New Zealand, Christchurch, Canterbury, New Zealand
- Poland (3):
  - Poland, Gdansk
  - Poland, Katowice
  - Poland, Lublin
- Spain (3):
  - Spain, Seville, Andalusia
  - Spain, Girona, Cataluyna
  - Spain, Madrid
- Ukraine (6):
  - Ukraine, Ivano-Frankivsk
  - Ukraine, Kharkiv
  - Ukraine, Odesa
  - Ukraine, Poltava
  - Ukraine, Ternopil
  - Ukraine, Vinnytsa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meng TC, Szaflarski JP, Chen L, Brunnert M, Campos R, Van Ess P, Pullman WE, Fakhoury T. Psychosocial outcomes of repeated treatment of seizure clusters with midazolam nasal spray: Results of a phase 3, open-label extension trial. Epilepsy Behav. 2023 Jan;138:108989. doi: 10.1016/j.yebeh.2022.108989. Epub 2022 Nov 18. PMID 36410152
- [Derived] Wheless JW, Meng TC, Van Ess PJ, Detyniecki K, Sequeira DJ, Pullman WE. Safety and efficacy of midazolam nasal spray in the outpatient treatment of patients with seizure clusters: An open-label extension trial. Epilepsia. 2019 Sep;60(9):1809-1819. doi: 10.1111/epi.16300. Epub 2019 Jul 29. PMID 31353457

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The participant flow refers to the enrolled population and includes participants who did not treat a seizure cluster episode.
Groups:
- USL261: 5 mg intranasal midazolam
  USL261
Period: Overall Study
Arm/Group | USL261
Started | 175 (Completed Study P261-401 and rolled over to Study P261-402)
Exposed | 161 (Treated at least 1 seizure cluster with USL261)
Completed | 1 (Completed under initial protocol duration of 2 years; amended protocol open-ended duration)
Not Completed | 174
Not completed — Discontinued prior to study treatment | 14
Not completed — Site closure | 62
Not completed — Study termination | 29
Not completed — Withdrawal by Subject | 25
Not completed — No treated SCs within protocol window | 13
Not completed — Noncompliance | 8
Not completed — Caregiver no longer available | 7
Not completed — Adverse Event | 4
Not completed — Protocol Violation | 4
Not completed — Lack of Efficacy | 4
Not completed — Investigator no longer available | 2
Not completed — Study drug not available | 2

BASELINE CHARACTERISTICS:
Population: Participants exposed to at least 1 dose of USL261
Arm/Group | USL261
Number analyzed (Participants) | 161
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 153
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 153
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Participant in Race unknown category reported race as "Slavic"
  Participants
    American Indian or Alaska Native | 2
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 4
    White | 152
    More than one race | 0
    Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  Canada | 1
  Hungary | 10
  United States | 56
  Ukraine | 53
  Poland | 12
  Israel | 5
  Australia | 12
  Germany | 7
  Spain | 5
Body Mass Index [Median (Full Range); unit: kg/m˄2] — Population: Height not reported for some participants
  kg/m˄2
    number analyzed (Participants) | 159
    (all) | 24.7 [17.7 to 43.0]
Seizure cluster episodes in year before Visit 1 in Study P261-401 [Median (Full Range); unit: seizure cluster episodes] | 18.0 [3 to 999]
Years had seizure cluster episodes prior to Study P261-401 [Median (Full Range); unit: years] — Population: Unknown or data entered as indefinite (eg >3) for some participants
  years
    number analyzed (Participants) | 157
    (all) | 5.00 [0.3 to 48.0]
Typical number of seizures in seizure cluster episode [Median (Full Range); unit: seizures] | 6.0 [2 to 170]
Typical duration of seizure cluster episode [Median (Full Range); unit: hours] — Population: Non-numerical duration (eg "several" hours) reported for some participants
  hours
    number analyzed (Participants) | 154
    (all) | 1.00 [0.0 to 72.0]

OUTCOME MEASURES:

1. Primary Outcome: Duration of Safety Observation
Description: Duration of participant study participation for collection of long term safety data
Time Frame: From Baseline/(Screening) to End of Safety-Follow-up (up to 56 months) as per assessment table of the study.
Population: Participants who received at least 1 dose of USL261 5mg on study
Measure: Median (Full Range); unit: months
Arm/Group | USL261
Number analyzed (Participants) | 161
months | 16.80 [1.0 to 55.7]

2. Primary Outcome: Participants Meeting Predefined Safety Criteria for Vital Signs
Description: Participants meeting predefined safety criteria for vital signs (systolic blood pressure [SBP] <85 mm Hg, SBP change from baseline >/= 40 mm Hg, diastolic BP [DBP] <50 mm Hg, DBP change from baseline >/=30 mm Hg, pulse rate <50 beats per minute (bpm), pulse rate >120 bpm, pulse rate change >/= 40 bpm at any visit post baseline or for caregiver recorded participant respiration rate [RR] <8 breaths per minute (brpm) or >24 brpm) after any USL261 treated seizure cluster episode. Abnormal vital signs were assessed separately by investigator and recorded as adverse events if applicable.
Time Frame: From Baseline/(Screening) to End of Safety-Follow-up (up to 56 months) as per assessment table of the study.
Population: Participants who received at least 1 dose of USL261 5 mg on study
Measure: Count of Participants; unit: Participants
Groups:
- USL261: USL261 5 mg or USL261 5 mg + 5 mg for a treated seizure cluster episode
Arm/Group | USL261
Number analyzed (Participants) | 161
Participants
  SBP <85 mm Hg | 0
  SBP change from baseline ≥ 40 mm Hg | 1
  DBP <50 mm Hg | 2
  DBP change from baseline ≥ 30 mm Hg | 3
  Pulse rate <50 bpm | 2
  Pulse rate >120 bpm | 1
  Pulse rate change from baseline >/= 40 bpm | 4
  Caregiver recorded RR <8 brpm | 1
  Caregiver recorded RR >24 brpm | 29

3. Primary Outcome: Participants With Laboratory Abnormalities Meeting Predefined Criteria
Description: Participants with abnormal laboratory finding, at any time post baseline, meeting predefined criteria. Abnormal laboratory findings were assessed separately by investigator and recorded as adverse events if applicable. Alanine aminotransferase (ALT); Alkaline phosphatase (ALP); Aspartate aminotransferase (AST); Gamma glutamyl transferase (GGT); upper limit of normal (ULN)
Time Frame: From Baseline/(Screening) to End of Safety-Follow-up (up to 56 months) as per assessment table of the study.
Population: Participants who received at least 1 dose of USL261 5 mg on study
Measure: Count of Participants; unit: Participants
Arm/Group | USL261
Number analyzed (Participants) | 161
Participants
  ALT >ULN & ≤3xULN | 26
  Albumin <30 g/L | 2
  ALP >2.5xULN | 1
  AST >ULN & ≤3xULN | 17
  AST >5x ULN & <20xULN | 1
  Bicarbonate <15.9 mmol/L | 6
  Cholesterol >7.75 mmol/L | 5
  Creatinine >1.5xULN | 1
  Creatinine >2x baseline | 2
  GGT >2.5xULN | 14
  Glucose <3 mmol/L | 3
  Glucose <8.9 mmol/L | 5
  Phosphate <0.8 mmol/L | 13
  Potassium >5.5 mmol/L | 5
  Sodium <130 mmol/L | 11
  Sodium >150 mmol/L | 1
  Hemoglobin <100 g/L | 5
  Hemoglobin decrease 20 g/L | 10
  Leukocytes <3x10^9/L | 4
  Lymphocytes <0.8x10^9/L | 4
  Neutrophils <1.5x10^9/L | 8

4. Primary Outcome: Participants With Clinically Significant Abnormalities Physical Examination
Description: Participants with abnormal findings, at any time post baseline, on physical examination considered clinically significant by the investigator.
Time Frame: From Baseline/(Screening) to End of Safety-Follow-up (up to 56 months) as per assessment table of the study.
Population: Participants who received at least 1 dose of USL261 5 mg on study
Measure: Count of Participants; unit: Participants
Arm/Group | USL261
Number analyzed (Participants) | 161
Participants
  Skin | 2
  Head/Eyes/Ears/Nose/Throat | 0
  Neck | 1
  Thyroid | 0
  Lungs | 0
  Heart | 0
  Abdomen | 0
  Lymph nodes | 0
  Extremities | 0

5. Primary Outcome: Participants With Clinically Significant Abnormalities on Neurologic Examination
Description: Participants with abnormal findings, at any time post baseline, on neurologic examination considered clinically significant by the investigator
Time Frame: From Baseline/(Screening) to End of Safety-Follow-up (up to 56 months) as per assessment table of the study.
Population: Participants who received at least 1 dose of USL261 5 mg on study
Measure: Count of Participants; unit: Participants
Arm/Group | USL261
Number analyzed (Participants) | 161
Participants
  Mental status | 10
  Cranial nerves II-XII | 1
  Motor strength of limbs | 2
  Deep tendon reflexes | 2
  Sensory exam | 1
  Station and gait | 5
  Hopping | 0
  Romberg test | 0
  Finger-to-nose test | 1
  Heel-to-shin test | 1
  Rapid alternating movements | 2
  Nystagmus | 0
  Tremor/Other abnormal movements | 0

6. Primary Outcome: Participants With Clinically Significant Abnormalities on Nasal Examination
Description: Participants with abnormal findings, at any time post baseline, on nasal examination considered clinically significant by the investigator
Time Frame: From Baseline/(Screening) to End of Safety-Follow-up (up to 56 months) as per assessment table of the study.
Population: Participants who received at least 1 dose of USL261 5 mg on study
Measure: Count of Participants; unit: Participants
Arm/Group | USL261
Number analyzed (Participants) | 161
Participants | 1

7. Primary Outcome: Participant Change in B-SIT Score
Description: Change in participant Brief Smell Identification Test (B-SIT) score from baseline to last visit with assessment. The B-SIT is a self-administered 12-item test; the score indicates odors correctly identified (0 to 12). The B-SIT was added while the study was already ongoing (Protocol Amendment 4, 20 May 2015) in response to a regulatory request. The test was only implemented at sites in the United States and included only participants considered by the investigator to have adequate cognitive ability to perform the test. Baseline was defined as the latest non-missing value prior to administration of USL261 in the Test Dose Phase of Study P261-401.
Time Frame: From Baseline/(Screening) to End of Safety-Follow-up (up to 56 months) as per assessment table of the study.
Population: Participants who received at least 1 dose of USL261 5 mg on study, had a baseline B-SIT in Study P261-401, and a post-baseline B-SIT in Study P261-402.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | USL261
Number analyzed (Participants) | 9
score on a scale | -0.6 (1.2)

8. Primary Outcome: Participants With Suicidal Ideation
Description: Participants with suicidal ideation reported on Columbia-Suicide Severity Rating Scale (C-SSRS) questionnaire at any post-baseline visit. Responses including: Wish to be Dead; Non-Specific Active Suicidal Thoughts; Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Active Suicidal Ideation with Specific Plan and Intent; and Any Suicidal Ideation Regardless of Type.
Time Frame: From Baseline/(Screening) to End of Safety-Follow-up (up to 56 months) as per assessment table of the study.
Population: Participants who received at least 1 dose of USL261 5 mg on study
Measure: Count of Participants; unit: Participants
Arm/Group | USL261
Number analyzed (Participants) | 161
Participants
  Wish to be dead | 3
  Non-specific active | 3
  Active without specific plan | 3
  Active with specific plan/intent | 1
  Any suicidal ideation | 4

9. Primary Outcome: Emergency Room/Emergency Medical Service Visits
Description: Participants requiring emergency room (ER)/emergency medical service (EMS) visit within 24 hours after any USL261 treated seizure cluster (including for continued seizures)
Time Frame: From Baseline/(Screening) to End of Safety-Follow-up (up to 56 months) as per assessment table of the study.
Population: Participants who received at least 1 dose of USL261 5 mg on study
Measure: Count of Participants; unit: Participants
Arm/Group | USL261
Number analyzed (Participants) | 161
Participants | 20

10. Secondary Outcome: Number of Treated Seizure Clusters Meeting Criteria for Treatment Success
Description: Number of Treated Seizure Clusters Meeting Criteria for Treatment Success: Termination of seizure(s) within 10 minutes and no recurrence within 6 hours after administration of first dose of USL261 (intranasal midazolam 5 mg)
Time Frame: 6 hours after first dose of USL261 for each treated seizure cluster
Population: Seizure cluster episodes treated with first dose of USL261
Measure: Count of Units; unit: Seizure cluster episodes
Units Other Than Participants: Seizure cluster episodes
Arm/Group | USL261
Number analyzed (Participants) | 161
Number analyzed (Seizure cluster episodes) | 1998
Seizure cluster episodes | 1108

ADVERSE EVENTS:
Time Frame: Original protocol - each participant 2 years from enrollment; Amended protocol - each participant open-ended from enrollment (up to 4 years or longer as approved by Health Authority where study being conducted). Actual individual participant duration 1.0 to 55.7 months.
Description: Adverse events collected at each visit from participant and/or caregiver. Due to intermittent treatment (qualifying seizure clusters), short systemic half-life of active (midazolam), and long participant duration, treatment emergent adverse event within 2 days after each treated seizure cluster are reported. Seizures were not considered adverse events unless worsening from underlying condition.
Arm/Group | USL261
All-Cause Mortality (participants affected / at risk) | 0/161
Serious Adverse Events (participants affected / at risk) | 8/161
Other Adverse Events (participants affected / at risk) | 33/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | USL261 (N=161)
Seizure cluster (Nervous system disorders) | 2 (4)
Convulsion (Nervous system disorders) | 2 (3)
Status epilepticus (Nervous system disorders) | 2 (2)
Epilepsy (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | USL261 (N=161)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 20 (96)
Somnolence (Nervous system disorders) | 15 (92)
Headache (Nervous system disorders) | 10 (27)

LIMITATIONS AND CAVEATS:
Open-label, non-comparative design. Potential participation bias due to participants and/or caregiver perceived efficacy/safety in prior study. Seizure data capture in diaries diminished over time in some participants due to length of study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A manuscript or abstract should not be submitted by investigator(s) for publication or presentation until a New Drug Application is approved by the US FDA or permission is granted in writing by sponsor.

DOCUMENTS (2):
  • Study Protocol (2015-05-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT01529034/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT01529034/SAP_001.pdf